CLINICAL TRIAL: NCT07132827
Title: A Multicentre, Randomised, Double-Blind, Placebo-Controlled, Parallel-Group Phase 3 Efficacy and Safety Study of SHR-1905 in Patiens With Chronic Rhinosinusitis With Nasal Polyps
Brief Title: Efficacy and Safety of SHR-1905 Injection in Subjects With Chronic Rhinosinusitis With Nasal Polyps
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1905-301
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-06

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1905 Injection (Experimental)
  Interventions: Drug: SHR-1905 Injection
- SHR-1905 Placebo Injection (Placebo Comparator)
  Interventions: Drug: SHR-1905 Placebo Injection

INTERVENTIONS:
Drug: SHR-1905 Injection — SHR-1905 Injection
  Arms: SHR-1905 Injection
Drug: SHR-1905 Placebo Injection — SHR-1905 Placebo Injection
  Arms: SHR-1905 Placebo Injection

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of SHR-1905 injection in subjects with chronic rhinosinusitis with nasal polyps (CRSwNP)

ELIGIBILITY:
Inclusion Criteria:

1. Weight ≥40kg
2. Diagnosed with chronic rhinosinusitis with nasal polyps (CRSwNP).
3. Bilateral nasal polyps at screening and baseline, total NPS ≥5, ≥2 points for each nostril.
4. NCS ≥2 at screening and baseline.
5. SNOT-22≥30 at screening period and baseline.
6. Recorded persistent NP symptoms for over 4 weeks prior to screening.
7. Subjects received standard therapy with intranasal corticosteroids (INCS) prior to randomization.
8. NP surgery in the past and/or SCS use within 1 years before screening(or with contraindications/ intolerances).

Exclusion Criteria:

1. Any comorbidities that may affect the efficacy evaluation of nasal polyps.
2. Any comorbidities except for asthma that may affect blood EOS levels.
3. Concomitant with immunodeficiency.
4. Concomitant with contraindications or not suitable for nasal endoscopy.
5. Uncontrolled hypertension and/or uncontrolled diabetes.
6. Concomitant with infection within 4 weeks prior to randomization.
7. Uncontrolled epistaxis within 4 weeks prior to randomization.
8. Major surgery performed within 3 months prior to randomization, or surgery planned during the study, or treatments that may affect evaluations according to investigators.
9. Parasitic infection within 6 months before randomization.
10. Sinus or intranasal surgery within 6 months prior to screening, or changes in the nasal walls caused by sinus or intranasal surgery that made NPS evaluation impossible.
11. Malignancies diagnosed within 5 years before randomization (except those with a low risk of metastasis or death).
12. Abnormalities of laboratory tests at screening or baseline.
13. Concomitant with active hepatitis B, positive hepatitis C virus antibodies, positive human immunodeficiency virus antibodies, or positive treponema pallidum antibodies.
14. Prolonged QTc interval or other clinically significant abnormal results of ECG at screening or baseline that may cause significant safety risks to subjects.
15. FEV1 before the use of bronchodilator (pre-BD) was less than 50% at screening.
16. Transfusion of blood products or immunoglobulin within 4 weeks prior to randomization.
17. SCS or additional INCS use within 4 weeks before randomization, or planned use during treatment period.
18. Regular use of decongestants (local or systemic) within 4 weeks before randomization, except for during the endoscopic procedure.
19. Adnimistration of live vaccine or viral vector vaccine within 4 weeks before randomization.
20. Allergen immunotherapy within 8 weeks before randomization.
21. Smoking at screening, or smoking cessation less than 6 months at screening.
22. Substance abuse, drug abuse, and/or excessive alcohol consumption within 1 year prior to randomization.

Pregnancy (including positive pregnancy test at screening or baseline), lactation, or pregnancy plan during study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Nasal polyp scores (NPS) | Baseline to Week 24
  Change from baseline in NPS at Week 24.
Nasal Congestion Scores (NCS) | Baseline to Week 24
  from baseline in NPS at Week 24.

SECONDARY OUTCOMES:
Lund Mackay score (LMK) from baseline on sinus CT scan | Baseline to Week 24
Loss of smell | Baseline to Week 24
Proportion of subjects with NPS≤1 point per nostril | Baseline to Week 24
Sino-nasal outcome test-22 (SNOT-22) scores | Baseline to Week 24
Total symptoms score (TSS) | Baseline to Week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & Ent Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided